CLINICAL TRIAL: NCT05023369
Title: Periarticular Administration of Dexamethasone to Improve Post-operative Pain, Function, Nausea, Hospitalization Length, and Risk of Complications in Patients Undergoing Hip Arthroplasty - A Randomized Trial
Brief Title: This is a Study to Verify if Periarticular Hip Injection of Corticosteroid After Hip Replacement Reduce the Pain and the Hospitalisation Time
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL - ORT - 028
Record Dates: First submitted 2021-08-12; First posted 2021-08-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone group (Experimental): Patient in this group will receive administration of 9 mg dexamethasone injected in the peri-articular tissues after the bone cut for hip endoprosthesis
  Interventions: Drug: Dexamethasone is a steroid drug and will be administered as an injectable solution (4mg/ml)
- Routine care (No Intervention): In this group only routinely performed anaesthesia protocol will be provided

INTERVENTIONS:
Drug: Dexamethasone is a steroid drug and will be administered as an injectable solution (4mg/ml) — Dexamethasone will be administered as an injectable solution (4mg/ml). Every ml of this solution contains 4 mg of dexamethasone sodium phosphate, corresponding to 3 mg of dexamethasone. Thus 3 ml of solution will be injected peri-articularly (arm-A)
  Other Names: Mephameson
  Arms: Dexamethasone group

SUMMARY:
The investigators are going to evaluate if periarticular corticosteroid injection during endoprothesis implantation can lead to any advantage to the patients, namely if it can reduce post-operative pain, lenght and cost of hospitalisation, use of analgesics drugs.

DETAILED DESCRIPTION:
Hip endoprothesis is a common orthopaedic prosthetic procedure, with continuously growing numbers in the last years, and the demand for this procedure is predicted to increase 4-fold by 2030. Recently, major interest has been given to improve postoperative pain management, to decrease the discomfort of the patients and with an outlook for reducing the length of hospital stay and decrease health-care costs. However, postoperative pain management is still problematic after this operation.

Post-operative pain control with the optimization of the analgesia protocol is a key aspect to be addressed to reduce the need for opioid analgesics, to quicken recovery and mobilisation, and to decrease the hospitalization length. To this regard, steroid supplementation is considered effective in decreasing post-operative pain. A recent meta-analysis from our research group on patients with total knee prosthesis proved the efficacy in decreasing post-operative pain. Moreover, a positive effect has been documented in terms of lower incidence of nausea and vomit, less post-operative range of motion limitation, and decreased systemic inflammatory response. All these benefits produced a shortened length of hospital stay without an increased risk of complications such as local infections.

Despite this overall positive effect of steroid supplementation, and their use by other specialties - e.g. anaesthesiology - and while there is now good evidence about the benefits of periarticular hip analgesic injection, e.g. FANS, opioid etc., there is still lacking evidence on the efficacy of periarticular corticosteroids in patients undergoing hip prosthetic replacement. In fact, there is a lack of information in the literature on their effectiveness in terms of pain management and function recovery. Furthermore, the influence of perioperative steroid application on the long-term follow-up results is poorly explored. This is a key issue, since the intensity of acute post-operative pain has been widely related to the risk of developing chronic post-operative pain, and thus the advantages of steroid supplementation, could go beyond the short-term pain relief and be even longer lasting.

This randomized controlled trial will thus investigate the benefit of implementing the peri-operative analgesia protocol not only to improve the acute post-operative recovery and shorten the hospital stay, but also to optimize the overall results after hip endoprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral cemented hip endoprosthesis for femoral neck fracture
* Patients aged 50-90 years old
* Patients with a BMI >18.5 and <35
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to steroids
* Revision endoprosthesis
* Active steroid or immunosuppressive therapy in the last 30 days before the operation
* Pregnant or breast-feeding women
* Presence of other clinically significant concomitant disease states (ASA IV)
* Uncontrolled diabetes mellitus
* Contraindications to NSAIDs
* Chronic systemic diseases as immunodeficiency, autoimmune disease (Systemic Lupus Erythematosus, SLE), gout, rheumatic arthritis
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 3 days after surgery
  The mean post-operative daily pain in the first three days after surgery assessed with the 0-10 numeric rating scale (NRS)

SECONDARY OUTCOMES:
Hip pain and function on a numeric rating scale (NRS) | Up to 24 months
  Hip pain and general function documented on a 0-10 NRS preoperatively and during the first 3 months, and reported on a 0-10 NRS at 2 and 6 weeks, 3, 6, 12, 24 months
Hip pain, function and quality of life on Harris Hip Score | Up to 24 months
  hip pain, function and quality of life evaluated by the validated clinical Harris Hip Score preoperatively and at 2 and 6 weeks, and at 3, 6, 12, 24 months postoperatively.
  The Harris Hip Score is a measure of dysfunction; the maximum score possible is 100 and the higher the score, the better the outcome for the individual.
Hip pain, function and quality of life on EQ-5D-5L Score | Up to 24 months
  hip pain, function and quality of life evaluated by the validated patient reported outcome measures EQ-5D-5L Scores preoperatively and at 2 and 6 weeks, and at 3, 6, 12, 24 months postoperatively
PainDETECT | Up to 24 months
  PainDETECT questionnaire for identifying neuropathic pain component and patient satisfaction on a two-level scale at 6, 12, 24 months
Nausea | 3 days after surgery
  Post-operative nausea documented during the 3 first post-operative days (both incidence and intensity on a 0-10 NRS)
Opioids and analgesic | Up to 24 months
  Post-operative opioids and analgesic drugs consumption documented with Medication Quantification Scale score (MQS) daily during the first 6 weeks and then at 3, 6, 12, 24 months postoperatively
PCR & ESR | 3 days after surgery
  Post-operative inflammatory response in terms of hematic C-Reactive Protein (CRP) and erythrocyte sedimentation rate (ESR) documented every day in the first 3 post-operative days
Mobilization | Up to week 2
  Time from surgery to first mobilization
Length of hospital stay | Up to week 2
  The length of hospital stay
Patient Satisfaction | reported on a 0-10 NRS at 2 and 6 weeks, 3, 6, 12, 24 months
  the satisfaction of the patient with the surgical procedure
Hip ROM | evaluation of range of motion preoperatively, at discharge and at 2 and 6 weeks, and at 3, 6, 12, 24 months postoperatively.
  range of movement of the operated hip

CONTACTS AND LOCATIONS:
Overall Officials: Christian MD Candrian, Prof., Principal Investigator — EOC
Locations (1):
- Christian Candrian, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No